CLINICAL TRIAL: NCT05330234
Title: Usability Study of OnTrack Tools: a Study to Assess the Usability of a Clinician-facing Software Application to Support Arm Rehabilitation After Stroke.
Brief Title: Usability Study of OnTrack Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22CX7578
Record Dates: First submitted 2022-04-01; First posted 2022-04-15 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Research With Clinical Staff in Stroke Rehabilitation
Keywords: stroke, rehabilitation, neurology, digital health
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This study aims to assess the usability of the OnTrack Tools GUI under simulation. The study follows up from a study of the OnTrack system that demonstrated the feasibility and acceptability of the patient-facing component of the system by stroke survivors and therapists. The design of this study was developed through a collaborative approach between the study researchers, patients, and front-line therapists. The OnTrack intervention is being developed by Imperial College, this usability study is part of the development process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapists (Other): Single arm study. Participants are members of the therapy team at Imperial College Healthcare NHS Trust's stroke wards.
  Interventions: Device: OnTrack Tools

INTERVENTIONS:
Device: OnTrack Tools — The intervention is the OnTrack Tools system consisting of a graphical user interface (GUI) used to manage patients who are users of the OnTrack rehabilitation system. Participants will be asked to complete clinical and non-clinical tasks in simulation using OnTrack Tools. The themes for the scenarios of use presented in each of the three phases are summarised below:
  Phase 1 - Account creation, system onboarding and general system navigation. Phase 2 - Individual patient management. Phase 3 - Content and data management.

SUMMARY:
Aims: Assess the usability of OnTrack Tools, a clinician facing interface to manage stroke survivors using the OnTrack rehabilitation system. Background: Arm disability is a common problem after stroke that can lead to loss of independence, it affects

~450,000 people in the UK. Repetitive activity is critical for recovery but research shows people can struggle with intensity and keeping track of progress. The OnTrack system being developed at Imperial College London is a potential solution to this problem. Intervention: The OnTrack system consists of two software applications, OnTrack App - used by patients, and OnTrack Tools - used by clinicians. OnTrack Tools pulls data generated by the OnTrack App and enables the monitoring of clients' arm activity, and management of goals and educational content. The software is used to inform selfmanagement coaching by helping therapists understand more about how and when patients use their affected arm between treatment sessions. Design and methods: This study will assess the usability of the OnTrack Tools component of the system. The study will recruit stroke therapists from Imperial College Healthcare NHS Trust to provide feedback on the experience and usability of OnTrack Tools' graphical user interface (GUI). The study will be divided into three progressive cycles of testing, feedback and iteration. Each cycle will see participants individually completing specific tasks related to system navigation and the management of patients under simulation. Participants will complete outcome measures and take part in focus groups. Researchers will analyse and use the feedback to improve the GUI ready for the next testing cycle. Patient and public involvement: The project team includes a PPIE group of stroke survivors who oversee the project and help us with public facing documentation. They are members of the research team and are reimbursed for their time and travel, according to INVOLVE guidance. Dissemination: Results of the study will be written-up for technical reporting and publication. Participants will be provided with a summary of results at the end of the study. The study team will be providing general updates on the progress of the study via their social media channels (e.g. Twitter @OnTrackRehab @ImperialIGHI @HelixCentre).

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years old or over) Occupational Therapists and Physiotherapists (Band 4 to Band 8) working in the stroke wards at ICHT.

Exclusion Criteria:

* No exclusion criteria has been defined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Darzi, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan for individual participant data to be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Therapists: Single arm study. Participants are members of the therapy team at Imperial College Healthcare NHS Trust's stroke wards.
  OnTrack Tools: The intervention is the OnTrack Tools system consisting of a graphical user interface (GUI) used to manage patients who are users of the OnTrack rehabilitation system. Participants will be asked to complete clinical and non-clinical tasks in simulation using OnTrack Tools. The themes for the scenarios of use presented in each of the three phases are summarised below:
  Phase 1 - Account creation, system onboarding and general system navigation. Phase 2 - Individual patient management. Phase 3 - Content and data management.
Period: Overall Study
Arm/Group | Therapists
Started | 10
Phase 1 | 10
Phase 2 | 9
Phase 3 | 6
Completed | 6
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Therapists
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale (Phase 1)
Description: In systems engineering, the system usability scale (SUS) is a simple, ten-item attitude Likert scale giving a global view of subjective assessments of usability. It was developed by John Brooke[1] at Digital Equipment Corporation in the UK in 1986 as a tool to be used in usability engineering of electronic office systems.
  The measure is scored on a 0-100 scale, a higher score means a better outcome.
Time Frame: Up to 60 days.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Therapists (Phase 1): Single arm study. Participants are members of the therapy team at Imperial College Healthcare NHS Trust's stroke wards.
  OnTrack Tools: The intervention is the OnTrack Tools system consisting of a graphical user interface (GUI) used to manage patients who are users of the OnTrack rehabilitation system. Participants will be asked to complete clinical and non-clinical tasks in simulation using OnTrack Tools. The themes for the scenarios of use presented in each of the three phases are summarised below:
  Phase 1 - Account creation, system onboarding and general system navigation. Phase 2 - Individual patient management. Phase 3 - Content and data management.
Arm/Group | Therapists (Phase 1)
Number analyzed (Participants) | 10
score on a scale | 73.3 [62.5 to 90]

2. Primary Outcome: System Usability Scale (Phase 2)
Description: as for outcome 1
Time Frame: Up to 60 days
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Therapists (Phase 2): Single arm study. Participants are members of the therapy team at Imperial College Healthcare NHS Trust's stroke wards.
  OnTrack Tools: The intervention is the OnTrack Tools system consisting of a graphical user interface (GUI) used to manage patients who are users of the OnTrack rehabilitation system. Participants will be asked to complete clinical and non-clinical tasks in simulation using OnTrack Tools. The themes for the scenarios of use presented in each of the three phases are summarised below:
  Phase 1 - Account creation, system onboarding and general system navigation. Phase 2 - Individual patient management. Phase 3 - Content and data management.
Arm/Group | Therapists (Phase 2)
Number analyzed (Participants) | 9
score on a scale | 78.3 [72.5 to 92.5]

3. Primary Outcome: System Usability Scale (Phase 3)
Description: as for outcome 1
Time Frame: Up to 60 days.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Therapists (Phase 3): Single arm study. Participants are members of the therapy team at Imperial College Healthcare NHS Trust's stroke wards.
  OnTrack Tools: The intervention is the OnTrack Tools system consisting of a graphical user interface (GUI) used to manage patients who are users of the OnTrack rehabilitation system. Participants will be asked to complete clinical and non-clinical tasks in simulation using OnTrack Tools. The themes for the scenarios of use presented in each of the three phases are summarised below:
  Phase 1 - Account creation, system onboarding and general system navigation. Phase 2 - Individual patient management. Phase 3 - Content and data management.
Arm/Group | Therapists (Phase 3)
Number analyzed (Participants) | 6
score on a scale | 77.1 [72.5 to 82.5]

4. Secondary Outcome: Post-Study System Usability Questionnaire (PSSUQ)
Description: The PSSUQ (Post-Study System Usability Questionnaire is a 16-item standardized questionnaire. It is widely used to measure users' perceived satisfaction of a website, software, system or product at the end of a study.
  PSSUQ follows a 7-point Likert Scale (+ NA option).
  1 is "strongly agree" and 7 is "strongly disagree"
  Results are calculated by averaging the scores from the 7 points of the scale.
  The PSSUQ has one overall score and 3 sub-scales, namely system usefulness, information quality, and interface quality scored as follows:
  Overall: the average scores of questions 1 to 16 System Usefulness (SYSUSE): the average scores of questions 1 to 6 Information Quality (INFOQUAL): the average scores of questions 7 to 12 Interface Quality (INTERQUAL): the average scores of questions 13 to 15
  The lower the scores, the better the performance and the higher the perceived satisfaction.
Time Frame: Up to 60 days.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Therapists (Phase 3)
Number analyzed (Participants) | 6
score on a scale
  Overall | 2.6 [1.7 to 3.1]
  SYSUSE | 2.5 [1.3 to 3.2]
  INFOQUAL | 2.7 [1.5 to 3.2]
  INTERQUAL | 2.6 [2 to 4]

ADVERSE EVENTS:
Time Frame: No adverse event data was collected for this study
Description: This was a simulation study involving staff members reviewing the interface of a software device
Arm/Group | Therapists
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT05330234/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT05330234/ICF_001.pdf